CLINICAL TRIAL: NCT00347282
Title: Post-enucleation Socket Syndrome Study (PESSS): Part 1 - Three Dimensional Volumetric Assessment of Anophthalmic Sockets With the New Multi-detector Computed Tomographic Technology
Brief Title: Post Enucleation Socket Syndrome Study
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Other Study IDs: R440/35/2005
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Eye Enucleation; Orbit Surgery; Postoperative Complications
Keywords: Post enucleation socket syndrome; Multi-slice computed tomography scan; Prospective studies; Tomography, X Ray Computed
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Superior sulcus deformity in post-enucleation socket syndrome (PESS) may pose a significant cosmetic blemish after enucleation surgery despite apparently adequate orbital volume replacement. The underlying reasons include the lack of accurate pre-operative volumetric assessment of the anophthalmic socket, leading to either under or over estimation of the orbital implant required and the shifting in orbital and periocular structures that may occur post enucleation. Conventional imaging studies (computed tomography and magnetic resonance imaging) have been used to study the anatomy of anophthalmic sockets, but there are several drawbacks such as poor image quality for detailed volumetric assessment, long exposure time with possible motion artifact and etc. The new multi-detector computed tomographic technology is the latest advance in diagnostic radiology that allows rapid high resolution images to be obtained for three dimensional reconstruction and volumetric assessment. This new imaging modality will contribute greatly to the understanding of PESS and the surgical planning of anophthalmic sockets reconstruction.

This is a pilot study aiming to collect clinical data on the volumetric and structural changes in PESS. The information obtained will:

1. allow more accurate volume estimation of the primary orbital implants prior to enucleation surgeries, thus minimize the development of PESS;
2. evaluate the volumetric & structural anomalies that constitute PESS
3. be used for the development of a new customized secondary orbital implant to manage superior sulcus deformity in PESS.

DETAILED DESCRIPTION:
Purpose:

Primary aim:

Three dimensional volumetric assessment of the changes in orbital soft tissues in patient with post-enucleation socket syndrome, using the new 16-slice multi-detector computed tomography scanner.

Background:

Post-enucleation socket syndrome (PESS - enophthalmos, superior sulcus deformity, ptosis or upper eyelid retraction and lower eyelid laxity1) is a well recognized late complication of enucleation surgery. The underlying pathophysiology, however, has not been well established. It is especially prominent when there is inadequate orbital volume replacement or contraction of the socket.2

Superior sulcus deformity (Fig.1) manifests as a deep groove or space between the upper eyelid and the superior orbital rim. In a review by Smerdon and Sutton, it was the only significant factor related to poor cosmetic satisfaction.3 It was suggested that the loss of orbital volume and relaxation of tissues were the causes.4

With the advance in orbital implant development, most patients received implant replacement during their enucleation surgery or shortly afterward to improve the cosmetic outcome. A survey among members of the American Society of Ophthalmic Plastic and Reconstructive Surgery reported a total of 2,779 primary orbital implant being performed in a year.5

An ideal orbital implant replaces 70-80% of the volume enucleated (~5ml, i.e. implant size 20-22mm), while the ocular prosthesis fills the rest (~2ml). But the predictions of implant size have been relatively subjective and inaccurate. They are influenced by factors like phthisis, configuration of the orbit, placement of the extraocular muscles, shape of the implant, the use of implant warps and the orbital fat volume.6 In a retrospective study by Kaltreider et al, 76% of the patients would benefit from a larger implant and 63% would need an implant size larger than 22mm.7 On the contrary, in a prospective study by Custer and Trinkaus, no implant of larger than 22mm was needed.8 However in both studies, patients with less volumetric replacement showed significantly more severe enophthalmos and superior sulcus deformity.

Different surgical procedures, mostly by secondary volume augmentation 9-19, have been suggested to treat superior sulcus deformity and PESS. They can be categorized into subperiosteal implants on the orbital floor or eyelid implants.20 Besides filling up the orbital volume, subperiosteal implants produce upward and forward displacement of orbital content to correct the superior sulcus deformity. Cosmetic improvement with the eyelid implants or filler material is achieved by adding bulk to the hollowed area below the brow and above the upper eyelid crease directly. In spite of these, information on accurate pre-operative volumetric assessment of the anophthalmic sockets remained inadequate, resulting in occasional revision of the volume augmented.21

Conventional imaging studies have been used for various oculoplastic conditions for more than two decades. In studying orbital anatomy and pathology, Nugent RA et al has demonstrated changes in the extraocular muscle (diameter & volume) in patients with Graves' orbitopathy with the second generation CT scanner and found to correlate well with the clinical findings22. In the area of anophthalmic sockets, both computed tomography (CT) and magnetic resonance imaging (MRI) have contributed to the understanding of the condition. With the use of high resolution CT, Smith et al had demonstrated deepening of the superior sulcus, sagging & retraction of the superior muscle complex, distal elevation & retraction of the inferior rectus and downward & forward redistribution of the orbital fat in 22 anophthalmic sockets without orbital implant insertion. They had further suggested a rotatory displacement of orbital content from superior to posterior and from posterior to inferior.23 In anophthalmic sockets with orbital implant, Detorakis's group had used 2mm cut MRI scan to demonstrate statistically insignificant decrease in rectus muscles volume and no change in orbital fat volume in 5 patients with enucleation surgery.24 Despite the information obtained, there were multiple drawbacks: poor image quality for detailed volumetric assessment, increased radiation exposure with separate scanning in axial and coronal planes, contra-indicated in patient with metallic foreign body injury, and long exposure time with possible motion artifact,25 and neither of the investigations have been translated into pre-operative volumetric assessment for surgical planning.

Multi-detector CT (MDCT) is the newest advance in CT technology. It provides unparalleled capabilities for detailed analysis of normal anatomy and pathology. MDCT allows very high resolution sub-millimeter image acquisition, and potentially true isotropic datasets, which is important in the production of good quality images on multi-planar reformation and volumetric assessment. In the study of anophthalmic sockets and PESS, high quality three dimensional reconstruction images mean accurate analysis of orbital soft tissue without the need of additional CT acquisition in a different plane. In a study comparing radiation exposure between MDCT and conventional CT in the imaging of para-nasal sinus, Zammit-Maempel et al have demonstrated an 84% reduction in radiation exposure with MDCT, the radiation dose of 9mGy was 54 times less than the threshold dose of 0.5-2Gy for detectable lens opacities26. Moreover, since the required coverage is less in the imaging of anophthalmic sockets, we can expect an even smaller and safer dose of radiation exposure. Last but not least, the 16-slice MDCT scanner is faster than conventional scanner, it can shorten the examination time and minimize motion artifact.

Despite all the published data, the patho-physiology of PESS remained unclear and the management of it is far from satisfactory. We are planning to answer some of the questions with anophthalmic sockets in 3 stages:

1. Anatomical and radiological analysis

   1. With this pilot study we are trying to identify the volumetric changes and the changes in anatomical relationship of the orbital soft tissue in anophthalmic sockets by comparing with contra-lateral eyes.
   2. Although MRI provide superior soft tissue contrast, CT still provides better detail of the eye, orbital soft tissue and bony orbit which is important for pre-operative surgical planning of secondary sub-periosteal orbital implant27.
2. Bioengineering and animal study (with the information obtained in part 1)

   1. We will assess the usefulness of MDCT in i. correct sizing of primary orbital implant in preventing PESS; and ii. correct sizing and effective placement of secondary orbital implant in restoring both the volumetric and positional changes in PESS.
   2. In addition, with the use of VGStudio MAX software, we may be able to offer customized secondary orbital implant for optimal correction of PESS.
3. Clinical trials

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent :

  * standard uncomplicated enucleation,
  * with primary hydroxyapatite or MEDPORE implant of size 20mm diameter or larger well placed within the posterior Tenon's space,
  * and re-suturing of the four recti muscles anterior to the equator,
* Aged 21 and above
* In good general health

Exclusion Criteria:

* Other types of orbital implant or implant size smaller than 20mm
* History of any disorders or surgery of the orbits: e.g. orbital trauma, repair of orbital fracture, orbital tumors, thyroid eye disease, orbital inflammatory disease, orbital irradiation
* History of any disorders or surgery of the extraocular muscles: e.g. myopathy, strabismus surgery
* History of any disorders or surgery of the eyelids: e.g. congenital ptosis, Horner's syndrome, ptosis surgery
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had enucleation surgery with primary orbital implant
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunny Shen, MBBS, MMed(Ophth), MRCS(Ed), Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

REFERENCES:
- [Background] Tyers AG, Collin JR. Orbital implants and post enucleation socket syndrome. Trans Ophthalmol Soc U K (1962). 1982 Apr;102 (Pt 1):90-2. No abstract available. PMID 6963069
- [Background] Smerdon DL, Sutton GA. Analysis of the factors involved in cosmetic failure following excision of the eye. Br J Ophthalmol. 1988 Oct;72(10):768-73. doi: 10.1136/bjo.72.10.768. PMID 3191079
- [Background] Bartlett RE. Plastic surgery for the enucleation patient. Am J Ophthalmol. 1966 Jan;61(1):68-78. doi: 10.1016/0002-9394(66)90749-5. No abstract available. PMID 5904380
- [Background] Su GW, Yen MT. Current trends in managing the anophthalmic socket after primary enucleation and evisceration. Ophthalmic Plast Reconstr Surg. 2004 Jul;20(4):274-80. doi: 10.1097/01.iop.0000129528.16938.1e. PMID 15266140
- [Background] Bilyk JR. Enucleation, evisceration, and sympathetic ophthalmia. Curr Opin Ophthalmol. 2000 Oct;11(5):372-86. doi: 10.1097/00055735-200010000-00015. PMID 11148706
- [Background] Kaltreider SA, Jacobs JL, Hughes MO. Predicting the ideal implant size before enucleation. Ophthalmic Plast Reconstr Surg. 1999 Jan;15(1):37-43. doi: 10.1097/00002341-199901000-00009. PMID 9949428
- [Background] Custer PL, Trinkaus KM. Volumetric determination of enucleation implant size. Am J Ophthalmol. 1999 Oct;128(4):489-94. doi: 10.1016/s0002-9394(99)00252-4. PMID 10577591
- [Background] Smith B, Obear M, Leone CR Jr. The correction of enophthalmos associated with anophthalmos by glass bead implantation. Am J Ophthalmol. 1967 Dec;64(6):1088-93. doi: 10.1016/0002-9394(67)93061-9. No abstract available. PMID 6072982
- [Background] Soll DB. Correction of the superior lid sulcus with subperiosteal implants. Arch Ophthalmol. 1971 Feb;85(2):188-90. doi: 10.1001/archopht.1971.00990050190012. No abstract available. PMID 5545718
- [Background] Iverson RE, Vistnes LM, Siegel RJ. Correction of enophthalmos in the anophthalmic orbit. Plast Reconstr Surg. 1973 May;51(5):545-54. doi: 10.1097/00006534-197305000-00010. No abstract available. PMID 4701236
- [Background] Hill JC, Radford CJ. Treatment of advancing enophthalmos in the ocular prosthetic patient: A preliminary report including a warning. Am J Ophthalmol. 1965 Sep;60(3):487-92. No abstract available. PMID 5825152
- [Background] Hneleski IS Jr, Shannon GM. Orbital floor implant. Am J Ophthalmol. 1973 Oct;76(4):540-2. doi: 10.1016/0002-9394(73)90745-9. No abstract available. PMID 4795524
- [Background] Spivey BE, Allen L, Stewart WB. Surgical correction of superior sulcus deformity occurring after enucleation. Am J Ophthalmol. 1976 Sep;82(3):365-70. doi: 10.1016/0002-9394(76)90485-2. PMID 786027
- [Background] Riebel O. Plastic surgery on the upper eye-lid after enucleation of the eye. Br J Ophthalmol. 1976 Oct;60(10):726-7. doi: 10.1136/bjo.60.10.726. No abstract available. PMID 1009045
- [Background] Smith B, Lisman RD. Use of sclera and liquid collagen in the camouflage of superior sulcus deformities. Ophthalmology. 1983 Mar;90(3):230-5. doi: 10.1016/s0161-6420(83)34569-3. PMID 6866445
- [Background] Leone CR Jr. Correction of superior sulcus defects after enucleation. Adv Ophthalmic Plast Reconstr Surg. 1990;8:209-13. PMID 2248712
- [Background] Soll DB. The anophthalmic socket. Ophthalmology. 1982 May;89(5):407-23. doi: 10.1016/s0161-6420(82)34774-0. PMID 7048182
- [Background] Nugent RA, Belkin RI, Neigel JM, Rootman J, Robertson WD, Spinelli J, Graeb DA. Graves orbitopathy: correlation of CT and clinical findings. Radiology. 1990 Dec;177(3):675-82. doi: 10.1148/radiology.177.3.2243967.
- [Background] Smit TJ, Koornneef L, Zonneveld FW, Groet E, Otto AJ. Computed tomography in the assessment of the postenucleation socket syndrome. Ophthalmology. 1990 Oct;97(10):1347-51. doi: 10.1016/s0161-6420(90)32411-9. PMID 2243686
- [Background] Detorakis ET, Engstrom RE, Straatsma BR, Demer JL. Functional anatomy of the anophthalmic socket: insights from magnetic resonance imaging. Invest Ophthalmol Vis Sci. 2003 Oct;44(10):4307-13. doi: 10.1167/iovs.03-0171. PMID 14507874
- [Background] De Potter P. Advances in imaging in oculoplastics. Curr Opin Ophthalmol. 2001 Oct;12(5):342-6. doi: 10.1097/00055735-200110000-00003. PMID 11588495
- [Background] Zammit-Maempel I, Chadwick CL, Willis SP. Radiation dose to the lens of eye and thyroid gland in paranasal sinus multislice CT. Br J Radiol. 2003 Jun;76(906):418-20. doi: 10.1259/bjr/82798696. PMID 12814929